CLINICAL TRIAL: NCT06141889
Title: A Phase 1, Single-dose, Open-label, Randomized Crossover and Multiple-dose, Open-label Study to Evaluate the Pharmacokinetics and Safety of Azelaprag in Older Adult Healthy Volunteers
Brief Title: Pharmacokinetics Study of Azelaprag (BGE-105) in Older Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioAge Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BGE-105-004
Record Dates: First submitted 2023-11-09; First posted 2023-11-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteer Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single dose, 2-way crossover in Part 1, then daily dosing for 14 days in Part 2 (Experimental): Study Part 1:
  Participants will receive a single Dose A or B on Day 1 and then followed by a crossover to a single Dose B or A on Day 8.
  Study Part 2:
  Participants in Study Part 2 will receive either a single Dose C or equivalent of Dose C administered twice daily, starting on Day 1 and through Day 14
  Interventions: Drug: Azelaprag

INTERVENTIONS:
Drug: Azelaprag — oral, apelin receptor (APJ) agonist
  Other Names: BGE-105

SUMMARY:
This study is a single-dose, open-label, randomized crossover and multiple-dose, open-label study to evaluate the PK of azelaprag in older adult healthy volunteers.

DETAILED DESCRIPTION:
This study is a single-dose, open-label, randomized crossover and multiple-dose, open-label study to evaluate the PK of azelaprag in older adult healthy volunteers. The study will enroll approximately 16 participants.

ELIGIBILITY:
Key Inclusion Criteria:

Patients who meet ALL the following inclusion criteria will be eligible to participate in the study:

1. Healthy male or female volunteers ≥ 60 years of age
2. No history or evidence of clinically relevant medical disorders
3. Body mass index (BMI) between 18 and 40 kg/m2
4. Acceptable physical examination findings, including vital signs, and electrocardiogram (ECG)
5. Acceptable clinical laboratory values
6. Female participants of non-childbearing potential

Key Exclusion Criteria:

1. Currently receiving treatment with another investigational drug or investigational device within 30 days (or 5 half-lives, whichever is longer)
2. Current or previous malignancy within 5 years, with the exception of non-melanoma skin cancers, cervical or breast ductal carcinoma in situ, or adenocarcinoma of the prostate
3. Positive test result for COVID (rapid test), human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or hepatitis C (HCV) antibodies
4. Use of any medications that might affect the metabolism of the study drug as assessed by the Investigator and Sponsor and use of any herbal supplements, vitamins, or nutritional supplements within the 14 days prior to the dose day of each dosing period or during study participation.
5. Planned elective surgery within 30 days prior to Screening, during the study period or before the participant's red blood cell (RBC) have returned to normal levels
6. Systolic blood pressure > 150 mm Hg or < 90 mm Hg or diastolic blood pressure > 95 mm Hg or < 60 mm Hg
7. Unwilling or unable to abstain from the use of nicotine or tobacco containing products (including but not limited to snuff, chewing tobacco, cigars, cigarettes, pipes, or nicotine patches) or the use of cannabis or marijuana
8. Positive urine drug screen or alcohol breath test at screening and/or known history of drug or alcohol abuse within 1 year prior to screening
9. History or evidence of any other clinically significant disorder, condition, or disease, that, in the opinion of the investigator or Sponsor medical monitor, if consulted, would pose a risk to participant safety, or interfere with the study evaluation, procedures, or completion
10. Concurrent or previous use of aspirin within 14 days and NSAIDs within 3 days before the dose day of each dosing period.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of azelaprag (BGE-105) after oral administration - AUC0-t | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, area under the curve (AUC) from time 0 to time of the last observed serum concentration (AUC0-t)
Pharmacokinetics of azelaprag (BGE-105) after multiple-dose (Part 2) - AUC0-24 | Study Part 2, Predose and post dose to 24 hours after the final dose is received.
  Assessment of PK parameter, area under the curve (AUC) over the dosing interval from time 0 to 24 hours following the final dose (AUC0-24)
Pharmacokinetics of azelaprag (BGE-105) after oral administration - AUC0-inf | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, UAC from time 0 to infinity (AUC0-inf)
Pharmacokinetics of azelaprag (BGE-105) after oral administration - Cmax | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, maximum observed serum concentration (Cmax)
Pharmacokinetics of azelaprag (BGE-105) after oral administration - Tmax | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, time to reach Cmax (Tmax)
Pharmacokinetics of azelaprag (BGE-105) after oral administration - T1/2 | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, terminal elimination half-life (T1/2)
Oral bioavailability of azelaprag after oral administration - Total body clearance | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, Total body clearance (CL)
Oral bioavailability of azelaprag after oral administration - Volume of distribution | Study Part 1, Predose and post dose to 144 hours after each dose received; Study Part 2, Predose and post dose to 96 hours after the final dose is received.
  Assessment of PK parameter, volume of distribution (Vz)

SECONDARY OUTCOMES:
Safety of azelaprag after oral administration - TEAEs | First dose to Day 21
  Number of participants with treatment emergent adverse events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Martin, MD, Study Director — BioAge Labs, Inc.
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No